CLINICAL TRIAL: NCT04653480
Title: Surufatinib and Toripalimab Combined With Chemotherapy for Second-line Treatment of Advanced RAS/BRAF Mutant and Microsatellite Stable Colorectal Cancer
Brief Title: Surufatinib, Toripalimab and Chemotherapy in Second-line MT and MSS CRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Director of Medical Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHRODITE
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — surufatinib; toripalimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib, Toripalimab and Chemotherapy (Experimental): Second line CRC patients received surufatinib 250mg po qd , toripalimab 3mg/kg ivgtt q2w and chemotherapy according to the first line treatment, until disease progression or intolerable toxicity
  Interventions: Drug: Surufatinib; Drug: Toripalimab; Drug: chemotherapy

INTERVENTIONS:
Drug: Surufatinib — 250mg per oral, once daily
Drug: Toripalimab — 3mg/kg IV, once every 2 weeks
Drug: chemotherapy — oxaliplatin or irinotecan based regimens, according to the first line treatment

SUMMARY:
To determine the efficacy and safety of surufatinib, toripalimab and chemotherapy in second-line RAS/BRAF mutant and MSS colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, ≤75 years
2. Histologically confirmed colorectal cancer with distant metastasis.
3. ECOG 0-1
4. Progression on first line therapy
5. RAS/BRAF mutant and microsatellite stable
6. Patients can swallow pills normally
7. Expected overall survival ≥6 months
8. Blood routine: no blood transfusion or blood products usage within 14 days, G-CSF or other hematopoietic stimulator was not used. WBC counts > 3000/µl，Absolute neutrophil count (ANC) ≥ 1500 cells/µl，Platelet count ≥ 100,000/µl，Hemoglobin ≥ 9.0 g/dL.
9. AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)，Serum bilirubin ≤ 1.5 x ULN，creatinine<ULN
10. Prothrombin time (PT), international standard ratio (INR) ≤1.5 × ULN
11. Patients who have not received immunotherapy
12. Women of childbearing age must be willing to use adequate contraceptives during the study period of drug treatment;
13. Informed consent has been signed.

Exclusion Criteria:

1. Patients have received ≥2 line systemic therapy;
2. Active bleeding within 3 months; Occurrence of arterial/venous thrombosis within 6 months; Hereditary or acquired bleeding (e.g., clotting dysfunction) or thrombotic tendencies; Full dose oral or injectable anticoagulants or thrombolytic drugs for therapeutic purposes are currently being used or have been used recently (10 days prior to the commencement of study treatment); Surgery (except for biopsy) was performed within 4 weeks prior to the study or the surgical incision was not fully healed; Aspirin (> 325 mg/ day) or dipyridamole, ticlopidine, clopidogrel, and silotazole are currently being used or have recently been used (10 days prior to the study).
3. Systemic corticosteroids or other systemic immunosuppressive drugs were used within 2 weeks prior to treatment. Immunosuppressive drugs were started or expected to be used during the trial. Inhaled corticosteroids, physiologic replacement doses of glucocorticoids are allowed.
4. Certain or suspected brain metastases.
5. The patient has a history of autoimmune disease.
6. Serious uncontrolled systemic diseases, such as severe active infections;
7. A person is known to be infected with the immunodeficiency virus (HIV) or known to be HIV-positive;
8. Patients have suffered from other malignancies in the past 5 years except cervical carcinoma in situ or basal cell carcinoma of the skin
9. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA >500 IU/mL) or active HCV carriers with HCV RNA can be detected. Remarks: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL) may be enrolled
10. Anti-infective therapy was not discontinued 14 days before the study;
11. A prior history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia, and symptomatic interstitial lung disease or the presence of active pneumonia on a chest CT scan within 4 weeks prior to the study.
12. Patients have a history of intestinal obstruction within six months. Patients with incomplete obstruction syndrome of ileus at the time of initial diagnosis may be enrolled in the study if they have received definitive (surgical) treatment to resolve the symptoms, as assessed by the investigator.
13. Patients Have high blood pressure that cannot be well controlled by antihypertensive medication (systolic ≥140 mmHg or diastolic ≥90 mmHg)
14. Urine routine indicated urinary protein ≥++ and confirmed 24-hour urinary protein >1.0g;
15. Known to be allergic to any study drug;
16. Patients have participated in other drug clinical studies within 4 weeks before enrollment;
17. Lactating women
18. According to the judgment of the researcher, the patient may have other factors that may affect the results of the study or cause the study to be terminated, such as alcohol abuse, drug abuse, other serious diseases (including mental diseases) requiring combined treatment. Patients have severe laboratory abnormalities, which will affect the safety of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 2 months
  the proportion of patients in a trial whose tumor is destroyed or significantly reduced by a drug. ORR is generally defined as the sum of complete responses (CRs) - patients with no detectable evidence of a tumor over a specified time period - and partial responses (PRs) - patients with a decrease in tumor size over a specified time period.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Refers to the time of death from enrollment to any cause
Progression Free Survival | 6 months
  the time elapsed between treatment initiation and tumor progression

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No